CLINICAL TRIAL: NCT06828471
Title: Social Cognition Training in Individuals With Huntington's Disease: A Feasibility Study
Brief Title: Social Cognition Training in Individuals With Huntington's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Samantha Patel, Assistant Professor in Neurological Sciences and Psychiatry and Behavioral Sciences, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24112605
Record Dates: First submitted 2025-02-11; First posted 2025-02-14 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Huntington's Disease (HD)
Keywords: Huntington's Disease; Social Cognition; Caregiver Burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social Cognition Training Group (Experimental)
  Interventions: Behavioral: Social Cognition Training

INTERVENTIONS:
Behavioral: Social Cognition Training — Neuroplasticity-based social cognition training that targets a range of social cognition skills, including visual and vocal affect perception, social cue perception, theory of mind, self-referential style, and empathy

SUMMARY:
Individuals with Huntington's Disease have impaired social cognition, which is the domain of cognition that allows individuals to understand others' perspectives so that they can navigate interpersonal actions successfully (e.g., understanding someone may be sad based of their facial emotion or tone of voice and then responding in a sympathetic manner). Impaired social cognition is associated with impaired social functioning, poor psychological wellbeing and increased caregiver burden, which is known to be significant among those who care for individuals with Huntington's Disease. Computerized social cognition training has been shown to improve social cognition in individuals with schizophrenia, who, like individuals with Huntington's disease, have cognitive impairments. The investigators propose a pilot study of computerized social cognition training in individuals with Huntington's disease. This will be a feasibility study that aims to show that social cognition training in HD can be studied in preparation for a larger randomized controlled trial. The investigators hypothesize that social cognition training can improve social cognition, social functioning, and quality of life in individuals with Huntington's Disease and decrease caregiver burden among those who care for individuals with Huntington's Disease.

ELIGIBILITY:
Inclusion Criteria for Individual with Huntington's Disease

* Diagnosed with Huntington's Disease based on genetic testing
* Must be between 18 and 65 years of age
* Native English speaker who is literate in English
* Stable psychotropic medication regimen for 4 weeks
* Must have a score of "somewhat easily" on all items in the CPQ-12
* MOCA >18
* Completed 12 years of schooling
* Access to laptop or mobile device
* Willingness to come in person 6-12 weeks after first visit

Inclusion Criteria for Caregiver of Individual with Huntington's Disease

* Lives with patient
* Must be between 18 and 65 years of age
* Native English speaker who is literate in English
* MOCA >26
* Willingness to come in person within 6-12 weeks after first visit

Exclusion Criteria for Individual with Huntington's Disease

* Any known neurological condition (other than Huntington's Disease).
* History of learning and/or intellectual disabilities
* Currently actively involved in any other interventional trial (i.e. have begun the intervention) or within 4 weeks of completing the final assessments of an interventional trial.
* Currently regularly completing a computerized cognitive training intervention.
* Active suicidal ideation with some intent

Exclusion Criteria for Caregiver of Individual with Huntington's Disease

* Inability to provide informed consent
* Active suicidal ideation with some intent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants willing to consider study out of those who have been approached | 32 months
Number of participants who adhered and completed the study | 32 months
Ease of program on a scale of 1 to 5 with 5 being "very easy." | 32 months
Participant satisfaction with the program | 32 months
  This will be a qualitative measure. The study staff will elicit from the participants what they liked about the program, what they did not like about the program, and what they would change about the program if they could.

SECONDARY OUTCOMES:
Change in accuracy on a facial emotion recognition task | 6-12 weeks
Change in accuracy on an empathic accuracy task | 6-12 weeks
  Participants view videos of individuals describing significant life events. Throughout the videos the participant are asked questions about the thoughts and feelings of the individual in the video.
Change in score on the Quality of Life in Neurological Disorders Ability to Participate in Social Roles and Activities (scores range from 45 to 225; higher score indicates better outcome) | 6-12 weeks
Change in score on the Quality of Life in Neurological Disorders Satisfaction with Social Roles and Activities Questionnaire (scores range from 45 to 225; higher score indicates better outcome) | 6-12 weeks
Change in score on the Quality of Life in Neurological Disorders Positive Affect and Wellbeing Questionnaire (scores range from 23 to 115; higher score indicates better outcome) | 6-12 weeks
Change in score on the Caregiver Burden Inventory (scores range from 0-96; lower score indicates better outcome) | 6-12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided